CLINICAL TRIAL: NCT01075633
Title: Colorectal Cancer Screening in Familiar-Risk Population: a Randomized Control Trial Comparing Immunochemical Fecal Occult Blood Testing Versus Colonoscopy
Brief Title: Colorectal Cancer Screening in Familiar-Risk Population: Immunochemical Fecal Occult Blood Testing Versus Colonoscopy
Acronym: COLONFAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Enrique Quintero (Other)
Responsible Party: Sponsor-Investigator, Enrique Quintero, PhD, Fundación Canaria Rafael Clavijo para la Investigación Biomédica
Organization: Fundación Canaria Rafael Clavijo para la Investigación Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COLONFAM
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Colorectal Cancer
Keywords: FOBT; colonoscopy; familiar risk; colorectal cancer; advanced adenoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fecal occult blood testing (Experimental): Immunochemical fecal occult blood test Annual (3 rounds), without diet restriction, 1 stool sample. Positive cut-off level: 50 ng/ml.
  Interventions: Procedure: Immunochemical fecal occult blood test And colonoscopy if test is positive
- Colonoscopy (Active Comparator): Colonoscopy with sedation.
  Interventions: Procedure: Colonoscopy with sedation

INTERVENTIONS:
Procedure: Immunochemical fecal occult blood test And colonoscopy if test is positive — Annual (3 rounds), without diet restriction, 1 stool sample. Positive cut-off level: 50 ng/ml.
  Arms: Fecal occult blood testing
Procedure: Colonoscopy with sedation — Colonoscopy with sedation
  Arms: Colonoscopy

SUMMARY:
This study is aimed: 1) to compare the accuracy of colonoscopy vs immunochemical faecal occult blood test (iFOBT) and colonoscopy when positive for colorectal cancer (CRC) screening in familiar-risk population and; 2) to determine the complications associated with both strategies.

DETAILED DESCRIPTION:
This is an observational, controlled, randomized phase III study to evaluate the effectiveness of the iFOBT for detecting advanced neoplasia (polyps > 1cm in size, high grade dysplasia or with villous component, or CRC) in first degree relatives of patients with CRC.

Index cases will be interviewed to obtain the family tree and their first-degree relatives will be contacted to invite them to participate in the study. Index-cases, will be randomized into one of the following two groups in order that their relatives receive the same screening strategy: A) colonoscopy; or B) annual iFOBT test (OC-Sensor®, cut off ≥50 ng/ml) and colonoscopy if positive. To determine the sensitivity and specificity of the iFOBT strategy, individuals randomized to group B will be invited to undergo a complete colonoscopy following two years follow-up. In addition, epidemiological data, personal history of disease, family history of neoplasm, characteristics of lesions at colonoscopy and histological diagnosis will be recorded.

To test the hypothesis of equivalence between the iFOBT test and colonoscopy for detecting advanced colorectal neoplasm, it was considered a probability of participation, detection capability and prevalence of advanced adenomas for iFOBT of 0.750, 0.565 and 0.077, respectively, being the product of them 0.033. In the case of colonoscopy, the likelihood of participation, detection capability and prevalence of advanced adenomas in this population at risk are 0,500, 0.965 and 0.077, respectively, and their product 0.037. Accordingly, for a Type I error (alpha) of 5%, a power of 80% and a maximum deviation between the probabilities of the two tests of 0.03 the number of subjects to be included per arm is 744

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 40-75 years, first degree relatives of patients with non-syndromic CRC

Exclusion Criteria:

* Personal history of CRC, colorectal adenoma, colorectal polyposis, or inflammatory bowel disease

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1501 (Actual)
Dates: Start 2006-01; Primary Completion 2011-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Advanced colorectal neoplasm detection rate [Time Frame: 2 years] [Designated as safety issue: No] | 2 years

SECONDARY OUTCOMES:
Complications rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Quintero, MD, Study Director — Fundación Canaria para la Investigación Biomédica Rafael Clavijo
Locations (1):
- Hospital Universitario de Canarias, Santa Cruz de Tenerife, Spain, Spain

REFERENCES:
- [Result] Gimeno-Garcia AZ, Quintero E, Nicolas-Perez D, Hernandez-Guerra M, Parra-Blanco A, Jimenez-Sosa A. Screening for familial colorectal cancer with a sensitive immunochemical fecal occult blood test: a pilot study. Eur J Gastroenterol Hepatol. 2009 Sep;21(9):1062-7. doi: 10.1097/MEG.0b013e3283293797. PMID 19307978
- [Derived] Quintero E, Carrillo M, Gimeno-Garcia AZ, Hernandez-Guerra M, Nicolas-Perez D, Alonso-Abreu I, Diez-Fuentes ML, Abraira V. Equivalency of fecal immunochemical tests and colonoscopy in familial colorectal cancer screening. Gastroenterology. 2014 Nov;147(5):1021-30.e1; quiz e16-7. doi: 10.1053/j.gastro.2014.08.004. Epub 2014 Aug 13. PMID 25127679